CLINICAL TRIAL: NCT03863041
Title: Study of Phosphorylated Metabolism Profile as Predictive Biomarker of Cognitive Decline in Memory Complaint.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRMAPHO
Record Dates: First submitted 2018-10-24; First posted 2019-03-05 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Memory Complaint; Alzheimer Disease; Phosphorylated Metabolism Profile; Magnetic Resonance Spectroscopy
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Additional MRI SCAN sequence (Other): Additional sequence performed during MRI scan
  Interventions: Other: Additional sequence performed during MRI scan

INTERVENTIONS:
Other: Additional sequence performed during MRI scan — An additional sequence will be performed during the MRI scan.

SUMMARY:
Alzheimer disease is a frequent disease in the late ages that results in global alteration of cognitive functions. In which memory complaint can be isolated in the early stages.

Physiopathology of neuronal degenerescence in Alzheimer disease is complex, two main histological lesions are known, amyloid plaques and neurofibrillar tangles. Beyond the histological knowledge, alterations of neuronal metabolism are described such as oxydative phosphorylation and glycolytic pathway. These metabolism alterations are involved in neuronal death.

Multi-nucleus magnetic resonance spectroscopy is a non-invasive non-irradiant imagery technique already used in routine. This technic allows the phosphoenergetic pool assessment, that inform about cellular metabolism.

The aim of the study is to explore the phosphorylated metabolism patterns as predictive biomarkers of cognitive decline in patients with a memory complaint diagnosed.

ELIGIBILITY:
Inclusion Criteria:

1. Memory complaint, leading to a medical visit at the Centre Mémoire de Ressources et de Recherche (CMRR) of Poitiers, and for which an MRI is needed in routine exploration.
2. Age inferior at 90 years old
3. Mini Mental State Examination (MMSE) score between 20 and 30
4. Patient without guardianship measure, without restricted liberty.
5. Patient who benefits from social security

Exclusion Criteria:

1. Vascular, tumor, inflammatory pathology diagnosed by MRI
2. Other diagnosed neurodegenerative disease than Alzheimer disease
3. Other non neurodegenerative neurological disease
4. Vital risk at short term
5. Severe and uncontrolled psychiatric disease

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
phosphorylated metabolism profile assessment as predictor of cognitive decline in patients with memory complaint. | ONE YEAR
  correlation between brain phosphorylated metabolism (Pcr, ATP, PME, PDE, cho, NAA, Cr, PH) at the inclusion and MMSE on 2 years.

SECONDARY OUTCOMES:
Correlation between phosphorylated metabolite and final diagnostic of Alzheimer disease or not. | ONE YEAR
  Correlation between brain metabolite (Pcr, ATP, PME, PDE, cho, NAA, Cr, PH) and Alzheimer disease final diagnostic.
Correlation between phosphoryled metabolite and variability of cerebro spinal fluid biomarkers | ONE YEAR
  Correlation between brain metabolite (Pcr, ATP, PME, PDE, cho, NAA, Cr, PH) and cerebro spinal fluid biomarkers (B-amyloid Tau protein and Phosphorylated-Tau Protein)
Correlation between multinuclear magnetic resonance spectroscopy data and severity of cognitive dysfunction, at the inclusion and at one year. | ONE YEAR
  Correlation between brain metabolite (Pcr, ATP, PME, PDE, cho, NAA, Cr, PH) and MMS score at the inclusion and at one year.
Evolution of multinuclear magnetic resonance spectroscopy data at one year and cognitive decline at one year. | ONE YEAR
  Comparison at the inclusion and at one year of brain metabolite (Pcr, ATP, PME, PDE, cho, NAA, Cr, PH) and MMS score.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU of Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No